CLINICAL TRIAL: NCT04954196
Title: Benefit of Amlodipine in HRT Cycle (Hormone Replacement Therapy) for Frozen Embryo Transfer in the Correction of Uterine Pulsatility Index: Randomized Controlled Double-blind Trial.
Brief Title: Benefit of Amlodipine in HRT Cycle for Frozen Embryo Transfer in the Correction of Uterine Pulsatility Index
Acronym: AMLODIP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL20_0092
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Frozen Embryo Transfer
Keywords: Frozen embryo transfer; Uterine artery pulsatility index; Implantation; Calcium channel blocker
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Amlodipine 5 mg capsules (Arrow Generics®) will be deblistered and repackaged in pill boxes of 28 capsules.
  Placebo capsules will be made of microcrystalline cellulose and will be identical in size and color to generic Amlodipine Arrow capsules. A mass uniformity check will be carried out. Placebo capsules will also be packaged in pill boxes of 28 capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amlodipine arm (Experimental): Single dose per os Amlodipine 5mg administration per day
  Interventions: Drug: Amlodipine 5mg
- Placebo arm (Placebo Comparator): Single dose per os placebo (microcrystalline cellulose) administration per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlodipine 5mg — HRT administration: On Day 1 of the cycle, HRT is planned in accordance with the department's standard practice.
  * The frozen embryo transfer will be performed 6 days after progesterone initiation.
  * The HRT will be maintained until the pregnancy test is performed: If the test is positive,HRT will be continued for up to 12 weeks of amenorrhea at the same doses and then gradually stopped. If the test is negative,HRT will be stopped gradually
  Amlodipine administration: On the day of the first monitoring Dm (corresponding to D13 D16 of the cycle), a single per os dose of amlodipine 5 mg is taken at night, neither the patient nor the investigator knows what drug is the patient getting. Monitoring is systematically performed the next morning.The treatment will be maintained until the pregnancy test is performed then if the test is positive, the treatment will be maintained for a total duration of 7 weeks.
  Other Names: AMLODIPINE ARROW GÉNÉRIQUES 5 mg
  Arms: Amlodipine arm
Drug: Placebo — HRT administration: On Day 1 of the cycle, HRT is planned in accordance with the department's standard practice.
  * The frozen embryo transfer will be performed 6 days after progesterone initiation.
  * The HRT will be maintained until the pregnancy test is performed: If the test is positive, HRT will be continued for up to 12 weeks of amenorrhea at the same doses and then gradually stopped. If the test is negative, HRT will be stopped gradually
  Placebo administration:On the day of the first monitoring Dm (corresponding to D13-D16 of the cycle), a single per os dose of placebo (Microcrystalline cellulose) is taken at night, neither the patient nor the investigator knows what drug is the patient getting. Monitoring is systematically performed the next morning.. The treatment will be maintained until the pregnancy test is performed, then if the test is positive, the treatment will be maintained for a total duration of 7 weeks.
  Arms: Placebo arm

SUMMARY:
Embryo implantation depends on two main factors: embryo grading quality and endometrial receptivity.Numerous tools have been suggested to evaluate these two factors. Measurement of the pulsatility index (PI) of the uterine arteries is associated with extremely low chances of pregnancy when it is high, especially higher than 3.

A pilot study of women with premature ovarian failure with at least one of the uterine PIs greater than 3 showed the efficiency of nifedipine in uterine vascularization. This calcium channel blocker, used sublingually in this study, significantly lowered uterine PI in nearly half an hour.

We are therefore interested in exploring this accessible, non-invasive and inexpensive tool, in the evaluation of endometrial receptivity before an embryo transfer.

DETAILED DESCRIPTION:
Embryo implantation is a key stage that depends on two main factors: embryo grading quality and endometrial receptivity. Numerous tools have been suggested to evaluate these two factors, without making it possible to predict with certainty the outcome of an embryo transfer in terms of pregnancy. However, some diagnostic tests have shown a good negative predictive value: it is the case of the measurement of the pulsatility index (PI) of the uterine arteries which is associated with extremely low chances of pregnancy when it is high, especially higher than 3 (Cacciatore et al., 1996; Steer et al., 1992).

The Pulsatility Index PI is calculated by the ratio between the maximum amplitude of the tracing and the mean velocity. It evolves according to downstream resistance. Uterine hypoperfusion would readily be associated with subfertility (Goswamy et al., 1988). The uterine arterial pulsatility index is easily accessible during pelvic ultrasound, with satisfactory intra- and inter-observer reproducibility (Steer et al., 1995). There is no significant difference between the measurement of the right and left uterine PI (Favre et al., 1993). Uterine PIs vary during the menstrual cycle (Goswamy and Steptoe, 1988) and depending on hormonal effects (de Ziegler et al., 1991; Strigini et al., 1995) or ovarian micropolycystic status (PCOS, syndrome of polycystic ovaries) of the patient (Resende et al., 2001). The impact of tobacco (Battaglia et al., 2011) and parity (Guedes-Martins et al., 2015) on uterine PIs is described in the literature. Age, although controversial, does not seem to have an impact on uterine PIs, at least in premenopausal women case (Check et al., 2000). Likewise, body mass index (BMI) could have an impact on PIs, as in increased PIs in obese women (Battaglia et al., 1996; Zeng et al., 2013) If high uterine PIs are associated with reduced chances of pregnancy, how can they be improved? A pilot study of women with premature ovarian failure with uterine PIs greater than 3 showed the efficiency of nifedipine in uterine vascularization. This calcium channel blocker, used sublingually in this study, significantly lowered uterine PI in nearly half an hour (Huissoud et al., 2004). This medication could therefore be promising in the treatment of patients in assisted medical reproduction (ART) for whom the measurements of the uterine PIs would be greater than 3 and therefore have lower chances of pregnancy.

This study aims to investigate weither the use of a calcium channel blocker (amlodipine) improves the value of uterine PIs in patients with at least one of the uterine PIs greater than 3, during a cycle for frozen embryo transfer (FET).

ELIGIBILITY:
Inclusion Criteria:

* Female subject
* 18 years (≤) age (≤) 38 years
* Patient scheduled for a blastocyst frozen transfer (vitrification on Day 5) on HRT cycle (hormone replacement therapy)
* Measurement of at least one of the two uterine PI (pulsatility index) greater than 3 (> 3) at the first monitoring Dm (corresponding to Day 13-Day 16 of the cycle)
* BMI ≤ 30 kg / m2
* Carrying out a transfer test qualified as easy (passage through the cervix of a flexible or rigid catheter, without anesthesia or Pozzi forceps)
* Collection and signature of free and informed consent
* Subject affiliated to or beneficiary of a health insurance plan

Exclusion Criteria:

* Active smoker patient (at least one cigarette a day at the enrollment in the study)
* Oocyte recipient patient
* A pre-implantation genetic screening (PGS) is planned for the patient
* Patient with stage 3 or 4 endometriosis, or adenomyosis
* Contraindication to the use of amlodipine (recent myocardial infarction less than one month old, severe angina pectoris, severe hepatic insufficiency, treatment with ciclosporin, hypotension, hypersensitivity to amlodipine, dihydropyridine derivatives)
* Concomitant use of inhibitors or enzyme inducers of CYP3A4
* Patient already being treated for high blood pressure
* Patient with an ovarian follicle recruitmant (> 12mm) during the first monitoring (the most conservative case)
* Patient participating in another human intervention study
* Patient in the exclusion period determined by a previous study
* Patient has already participated in this study
* Patient under legal protection, guardianship or curatorship
* Impossibility to give the patient clarifying information
* Impossibility to perform monitoring by an experienced sonographer
* Breastfeeding patient according to article L1121-5 of the CSP
* Patient protected or unable to give consent according to article L1121-8 of the Public Health Code (CSP)
* Vulnerable person according to article L1121-6 of the CSP

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patient scheduled for a blastocyst frozen transfer on HRT cycle
Enrollment: 0 (Actual)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2023-10-08 (Estimated); Study Completion 2024-09-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with 2 PI less then 3 Vs number of patients who performed ultrasound | seven days after initiation of treatment: Dm+7
  Compare the rate of patients with two PIs on Dm + 7 (corresponding to D20-23 of the cycle) less than 3 out of the number of patients who performed the Doppler ultrasound in both arms.

SECONDARY OUTCOMES:
Number of clinical pregnancies VS number of embryo transfers | 6 to 8 weeks after embryo transfer
  Compare the rate of embryo transfers performed vs the rate of clinical pregnancies in both arms.
  Clinical pregnancy is defined as pregnancy diagnosed by ultrasound with at least one gestational sac. Neither ectopic pregnancy nor pregnancy of undetermined location are considered to be pregnancy. This endpoint is measured by an independent blinded sonographer
number of miscarriages Vs number of embryo transfers | before 20 weeks of menorrhea
  Compare the rate of embryo transfers performed vs the rate of miscariages in both arms Miscarriage is defined as the loss of a clinical intrauterine pregnancy before 20 weeks of amenorrhea, confirmed by ultrasound
Number of live births Vs number of embryo transfers | Delivery time starting 20 weeks of amenorrhea
  Compare the rate of embryo transfers performed vs the rate of live births in both arms Live birth is defined as the birth after 20 weeks of at least one child born alive. The birth of twins or more is counted as a live birth.

CONTACTS AND LOCATIONS:
Overall Officials: Noémie RANISAVLJEVIC, MD, Study Director — Arnaud de Villeneuve University Hospital, Montpellier